CLINICAL TRIAL: NCT02838654
Title: Reliability of Epidural Waveform Analysis for Cervical Epidural Blocks
Brief Title: Cervical Epidural Waveform Analysis Using Pressure Monitoring Kit
Status: Completed | Type: Observational
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, associate professor, Keimyung University Dongsan Medical Center
Other Study IDs: 2016-05-037
Record Dates: First submitted 2016-07-12; First posted 2016-07-20 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Analysis, Event History
Keywords: cervical epidural space; wave form analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cervical epidural injection group: cervical epidural injection group
  Interventions: Procedure: cervical epidural injection

INTERVENTIONS:
Procedure: cervical epidural injection — sensitivity, specificity, positive predictive value, negative predictive value

SUMMARY:
The purpose of this study is to analyze the reliability of epidural wave form during cerivical epidural injection.

DETAILED DESCRIPTION:
The epidural space can be confirmed by loss of resistance (LOR) technique. However, LOR has very low specificity, although its sensitivity is high. Especially, cysts between ligaments, clefts in ligamentum flavum, paraspinal muscle and nonspecific spaces between muscles make false LOR.

Epidural wave form analysis (EWA) is very simple and reliable method which can substitue the LOR technique. If the epidural needle is located correctly in the epidural space, the investigators can observe a pulsatile wave and this pulsatile wave corresponds to arterial wave. Generally, sensitivity of EWA through needle is known to be superior to the sensitivity of EWA through catheter and most studies were focused on catheter EWA.

Cervical epidural space shows high false LOR rate and Lee et al demonstrated that false LOR at cervical epidural space was 68.7%. Therefore, nonspecificity of LOR technique require substitution method which can confirm epidural space.

ELIGIBILITY:
Inclusion Criteria:

* Cerivical Herniated nucleusus
* Cerivical spinal stenosis
* acute herpes zoster

Exclusion Criteria:

* Coagulopathy
* Infectious cervical disease
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who complain chronic neck pain due to cervical spinal disease or acute herpes zoster
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
epidural wave form reliability (sensitivity, specificity) analysis | 1 minute after the completion of the epidural injection

CONTACTS AND LOCATIONS:
Overall Officials: JiHEE Hong, MD, PhD, Principal Investigator — Keimyung University

IPD SHARING:
Plan to Share IPD: No